CLINICAL TRIAL: NCT01303042
Title: Multicenter Trial on Clinical Utility of Insulin Lispro Mix 50/50 T.I.D. Therapy in Patients With Type 2 Diabetes Mellitus
Brief Title: Efficacy of Insulin Lispro Mix 50/50 Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aichi Gakuin University (Other)
Responsible Party: Takahiro Tosaki, Aichi Gakuin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGU-247
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: insulin LISPRO; Insulin therapy; hemoglobin A1c protein, human; Blood Glucose Self-Monitoring; Quality of Life; Hypoglycemia; Diabetes Mellitus; 1,5-Anhydroglucitol
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypoglycemia; Diabetes Mellitus | interventions — isophane insulin, insulin lispro drug combination 50:50; insulin lispro, isophane insulin lispro drug combination (25:75)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulin lispro mix 50/50 (Experimental)
  Interventions: Drug: Insulin lispro mix 50/50

INTERVENTIONS:
Drug: Insulin lispro mix 50/50 — Insulin lispro mix 50/50 t.i.d : six months
  Other Names: Humalog Mix 50/50

SUMMARY:
Insulin therapy with lispro mix 50/50 t.i.d. is a treatment with a single insulin device. The management is comparatively simple and easy, but the curative effect is promising. It is also reported that noninferiority has been observed between basal/bolus therapy (BBT) and prandial premixed therapy (PPT, lispro mix 50/50 t.i.d.).

The purpose of this study is to evaluate whether change of insulin therapy from BBT (long-acting insulin at bedtime plus mealtime rapid-acting insulin) or analog insulin therapy t.i.d. (including therapies with aspart mix 70/30 and lispro mix 75/25) to lispro mix 50/50 t.i.d. improves glycemic control of patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Patients will continue existing insulin therapy for three months. After that, the investigators will change insulin therapy according to the insulin regimen below and continue the therapy for six months.

Patients will terminate from sulfonylurea treatment at the change of insulin therapy. The investigators will not change other oral hypoglycemic agents during the whole study period.

Regimen: Divide the total units of all insulin per day by three and equally apply the amount to mealtime injections of insulin lispro mix 50/50 t.i.d. When the unit is indivisible and the remainder is one unit, add it to the mealtime injection of breakfast. When the remainder is two units, add each unit to mealtime injections of breakfast and dinner.

Patients will terminate from the trial when their HbA1c increases by 1% and stays at the level for more than three months after the change of insulin regimen.

When there is a risk of hypoglycemia at the change of insulin regimen, the investigators will divide ninety percent of the total insulin units per day by three and equally apply the amount to mealtime injections of insulin lispro 50/50. When considered to be safe, the investigators will increase the insulin unit per day to the total insulin unit at the previous treatment within two months.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes patients who are treated with insulin basal/bolus therapy ( long-acting insulin at bedtime and mealtime rapid-acting insulin ) or analog insulin therapy t.i.d. (including therapies with aspart mix 70/30 and lispro mix 75/25) and whose HbA1c is above 7.4%.

Exclusion Criteria:

* Patients with renal failure with serum creatinine level ≧ 2.0
* Patients with hepatocirrhosis
* Patients with proliferative diabetic retinopathy or worse
* Patients with acute infectious disease
* Patients who are treated with steroids
* Patients with cancer
* Pregnant patients
* Patients who are decided to be inappropriate subjects by study physicians

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
pre- and postprandial glucose levels in SMBG | nine months

SECONDARY OUTCOMES:
Total score of Questionnaire on QOL | nine months
  Secondary end points include change in HbA1c and rates of hypoglycemia.

CONTACTS AND LOCATIONS:
Overall Officials: Takahiro Tosaki, MD, PhD, Study Chair — Dept. of Intern. Med., School of Dentistry, Aichi Gakuin University
Locations (4):
- Japan (4):
  - Dept. of Intern. Med., School of Dentistry, Aichi Gakuin University, Nagoya, Aichi-ken
  - Tosaki Clinic for Diabetes and Endocrinology, Nagoya, Aichi-ken
  - Diabetes Clinic, Okazaki East Hospital, Okazaki, Aichi-ken
  - Diabetes Center, Yokkaichi Social Insurance Hospital, Yokkaichi, Mie-ken